CLINICAL TRIAL: NCT07323810
Title: Monitoring the Effect of Mental Fatigue on Physical Performance Using Wearable Sensors and Physiological Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Bart Roelands, Professor Doctor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EC-2025-113
Record Dates: First submitted 2025-08-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Mental Fatigue
Keywords: Fatigue; Performance; Physiology; Wearables
MeSH Terms: conditions — Mental Fatigue; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Fatigue Condition (Experimental): The mental fatigue task will involve a modified Stroop test, adapted from previous research. Words will appear on the screen in 34-point font for 1000 milliseconds, with the inter-stimulus interval personalized based on each participant's Stroop max test performance. Stroop task duration will be 60 minutes for every participant. Participants will be instructed to respond as quickly and accurately as possible.
  Interventions: Behavioral: Mental Fatigue
- Control condition (No Intervention): The control task will consist of watching a pre-approved, emotionally neutral 60-minute documentary.

INTERVENTIONS:
Behavioral: Mental Fatigue — Mental fatigue (MF) is a psychobiological state characterized by feelings of tiredness and/or a measurable decline in performance following prolonged or intense cognitive activity.
  Arms: Mental Fatigue Condition

SUMMARY:
Mental fatigue (MF) negatively affects both cognitive and physical performance, increasing the risk of errors in high-stakes environments such as sports and surgery. Traditional methods to assess MF rely on subjective self-report scales, which are prone to bias, or on complex brain measurements (e.g. EEG) that are impractical outside laboratory settings. This study aims to develop a real-time, objective monitoring method for MF using wearable physiological sensors. The study will recruit healthy, trained runners (18-35 years old) who will complete both an MF-inducing cognitive task (Stroop test) and a control condition (watching a documentary) in a randomized, counterbalanced, crossover design. Heart rate variability, respiration rate, and pupil metrics will be continuously recorded using wearable devices. Machine learning models will be used to predict MF-level as well as the effect of MF on physical performance (5-km time trial on a treadmill) using the physiological data as input.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no neurological, cardiovascular or musculoskeletal disorders of any kind)
* Male or female
* No prior knowledge of the concept of MF
* No medication
* Non-smoker
* 18-35 years of age
* Experienced runners: (≥15km/week and/or ≥2u/week during the last 6 months)

Exclusion Criteria:

* Injuries in the past 6 months, affecting running performance
* Suffering from a chronic health condition (could be neurological, cardiovascular, internal or musculoskeletal)
* Participating in any concomitant care or research trials
* History of suffering from any mental/psychiatric disorders
* Use of medication
* Use of caffeine and heavy efforts 24 hours prior each trial
* Suffering from colour vision deficiencies
* Not eating a standardized meal, the morning of each trial and the evening before each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability time-domain parameters | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Root mean square of successive differences [RMSSD], standard deviation of normal-to-normal intervals [SDNN] in milliseconds.
Heart rate variability frequency-domain parameters | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Low-frequency (LF), High-frequency (HF) in milliseconds squared (ms²) and Low/high-frequency ratio [LF/HF]
Respiration rate | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Respiration rate (RR) will be measured as the number of breaths per minute (breaths/min)
Pupil diameter | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Pupil diameter (PD) will be measured in millimeters (mm) as an index of autonomic nervous system activity.
Blinking rate | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Blinking rate (BR) will be measured as the number of spontaneous blinks per minute (blinks/min)
Eyelid opening | Continuously during the cognitive intervention and control condition on the study day (approximately 75 minutes).
  Eyelid opening (EO) will be measured as the vertical distance between the upper and lower eyelid in millimeters (mm).
Cognitive Performance Accuracy | At baseline (pre-intervention), during the 60-minute cognitive intervention, and immediately after completion of the intervention on the study day (approximately 70 minutes total).
  Cognitive performance will be evaluated using a Go/No-Go task. The task begins with a general instruction screen, followed by the simultaneous presentation of two types of stimuli: a Go or No-Go signal and a left or right directional indicator. This results in four possible combinations: GoRight, GoLeft, NoGoRight, and NoGoLeft. When a Go signal appears, participants must respond by pressing the arrow key corresponding to the left or right direction. In contrast, when a No-Go signal is displayed, participants must withhold any response, regardless of the directional cue. This paradigm is designed to assess attention, response inhibition, working memory, and executive functions, all of which are known to be negatively affected by MF. Accuracy in percentage (%) of correct answers on this Go/No-Go task as well as accuracy during the Stroop intervention task will be measured.
Cognitive Performance Reaction Time | At baseline (pre-intervention), during the 60-minute cognitive intervention, and immediately after completion of the intervention on the study day (approximately 70 minutes total).
  Cognitive performance will be evaluated using a Go/No-Go task. The task begins with a general instruction screen, followed by the simultaneous presentation of two types of stimuli: a Go or No-Go signal and a left or right directional indicator. This results in four possible combinations: GoRight, GoLeft, NoGoRight, and NoGoLeft. When a Go signal appears, participants must respond by pressing the arrow key corresponding to the left or right direction. In contrast, when a No-Go signal is displayed, participants must withhold any response, regardless of the directional cue. This paradigm is designed to assess attention, response inhibition, working memory, and executive functions, all of which are known to be negatively affected by MF. Reaction time (RT) will be measured in milliseconds (ms) as the latency between stimulus onset and the participant's behavioral response (button press) on the Go/No-Go task and during the Stroop intervention task.
Physical performance: Time to Completion | Immediately after completion of the 60-minute cognitive intervention, during a single 5-km treadmill time trial on the study day (approximately 20 minutes).
  Participants will perform a 5-km running time trial on a treadmill to assess endurance performance under MF. The treadmill will be set at a 1% gradient, following established protocols to replicate outdoor running conditions. Before beginning the time trial, participants will complete a standardized warm-up for 5 minutes. To maintain self-paced running conditions, participants will receive real-time feedback on the distance covered but will not be provided with information about running speed or elapsed time. Researchers will remain present but will not offer verbal encouragement or pacing cues to ensure that the effort remains internally regulated. Once the 5-km distance is completed, participants will immediately stop running and step onto the treadmill's side platforms. The total time elapsed will be recorded.

SECONDARY OUTCOMES:
Subjective feeling of Mental Fatigue | At baseline (pre-intervention), every 5 minutes during the 60-minute cognitive intervention, and immediately after completion of the intervention on the study day.
  The Mental Fatigue Visual Annalogue Scale (0-10cm) will assess how mentally fatigued the participant is feeling (100 point VAS scale), and ranges from 'not at all' to 'completely exhausted'.
Mood | At baseline, prior to the start of each experimental and control trial on the study day.
  The Brunel Mood Scale (BRUMS) will be used to indicate mood, and serve as a control measure for both arousal as well as boredom. It features 24 mood descriptors (divided into 6 subscales (i.e. anger, confusion, depression, fatigue, tension and vigor)), where participants have to give a value for every mood on a 5-point Likert scale (i.e. 0=not at all to 4 = extremely) responding to the question: "how do you feel right now?"
Motivation | At baseline (pre-intervention) and immediately after completion of the 60-minute cognitive intervention on the study day.
  Moti-VAS: Motivation will be assessed using a VAS. Participants will be asked "How motivated do you feel for the upcoming task", and will be instructed to rate their answer on a 10cm line, with the statements "not at all" and "extremely motivated" at opposite ends of this line.
Sleepiness | At baseline (pre-intervention) and immediately after completion of the 60-minute cognitive intervention on the study day.
  The Karolinska Sleepiness Scale (KSS) will be conducted. This 10-point scale measures the subjective level of sleepiness and goes from 1 = 'extremely alert' to 10 = 'extremely sleepy, falls asleep all the time'.
Physical fatigue | Immediately prior to the physical performance test on the study day.
  To measure subjective feeling of physical fatigue, a P-VAS scale (0-10 cm) will be administered before each physical performance test to check the level of subjective physical fatigue of the participants. Participants will be asked to rate their general physical fatigue on a 10 cm line ranging from "not at all" to "completely exhausted".
Perceived physical exertion | During the 5-km treadmill time trial, assessed at the end of each kilometer on the study day.
  Rating of Perceived Exertion (RPE) will be measured using the Borg CR100® scale, which ranges from 0 to 100, with 0 representing "no exertion at all" and 100 representing "maximal exertion". Higher scores indicate greater perceived effort. Participants will be asked to provide an RPE rating at the end of each kilometre during the 5-km time trial.
Pacing | During the 5-km treadmill time trial, assessed at the end of each kilometer on the study day.
  Pacing will be assessed as the pattern of speed regulation across the 5-km time trial. Running speed (km/h) will be recorded continuously and summarized per kilometre to characterize pacing strategy (positive, negative, or even pacing). Relative speed will also be expressed as a percentage of average trial speed. Alongside total completion time, pacing will serve as an indicator of how participants distribute effort under self-paced running conditions.
  Participants will be asked every kilometer how fast they think they are running at that moment to verify any discrepancies with their actual running speed and observe whether there is a learning or condition effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels Labo voor Inspanning en Topsport, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No